CLINICAL TRIAL: NCT00268918
Title: A Phase I Trial of Docetaxel and PTK787 in Metastatic Breast Cancer Patients and Recurrent or Refractory Gynecological Cancer Patients
Brief Title: Docetaxel and PTK787 in Metastatic Breast Cancer Patients and Gynecological Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Susana M. Campos, MD, Medical Oncologist, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-020
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Cervical Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Breast Cancer
Keywords: PTK787; Metastatic breast cancer; Refractory gynecological cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Fallopian Tube Neoplasms; Breast Neoplasms | interventions — Docetaxel; vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel / PTK787 (Experimental): Docetaxel: Lead In: Given intravenously on Day 1 and Day 14 Afer Lead in: Given intravenously on day 1, 8, 15, 22 of each 28-day cycle.
  PTK787: Lead In: Given orally on day 4 and day 14 After Lead In: Given orally once a day.
  Interventions: Drug: Docetaxel; Drug: PTK787

INTERVENTIONS:
Drug: Docetaxel — Participants may continue receiving study drug as long as their disease does not worsen
  Other Names: Taxotere
Drug: PTK787 — Participants may continue receiving study drug as long as their disease does not worsen
  Other Names: Vatalanib

SUMMARY:
The main purpose of this study is to see if the study drug, PTK787, is safe and to find the highest dose that can be given safely without causing serious side effects.

DETAILED DESCRIPTION:
* Patients will come to the clinic once a week to receive study treatment. To help reduce the chance of an allergic reaction patients will take Decadron tablets orally the night before, the morning of and the evening of receiving chemotherapy.
* The lead-in schedule of dosing is as follows: Day 1: Taxotere intravenously; Day 4: PTK787 orally; Day 14: Taxotere and PTK787.
* After the lead-in schedule, a cycle will consist of 28 days. PTK787 will be given orally once a day without interruption. Taxotere will be given on Day 1, Day 8, Day 15 and Day 22.
* Before each dose of Taxotere, blood tests, urine tests, and a physical exam will be done. A radiological evaluation will be done every two months. If the patients tumor remains stable or shrinks in size, they may continue to stay on the study.
* Patients should not eat grapefruit or drink grapefruit juice during this study.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent gynecological cancers or metastatic breast cancer. Initial diagnosis must be confirmed histologically.
* Measurable disease or nonmeasurable disease
* Age > 18 years
* ECOG performance 0,1,2
* 4 weeks or greater since major surgery, 3 weeks or greater since chemotherapy
* Certain lab values
* Negative for proteinuria

Exclusion Criteria:

* Four or more treatment regimens
* History or presence of uncontrolled CNS disease
* Prior biologic or immunotherapies less than 3 weeks prior to registration
* Prior full field radiotherapy less than 4 weeks or limited field radiotherapy less than 2 weeks prior to registration
* Prior therapy with anti-VEGF agents
* Peripheral neuropathy with functional impairment > CTC grade 2
* Pregnant or breast feeding
* Concurrent severe and/or uncontrolled medical condition
* Chronic renal disease
* Acute or chronic liver disease
* Impairment of gastrointestinal function or GI disease
* Confirmed diagnosis of HIV infection are excluded at the investigators discretion
* Therapeutic warfarin sodium or similar oral anticoagulants that are metabolized by the cytochrome p450 system.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and the dose limiting toxicity of weekly Taxotere patients treated with PTK787. | 2 years

SECONDARY OUTCOMES:
To estimate the preliminary efficacy of this combination in both metastatic breast cancer patients and refractory gynecological patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susana M. Campos, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts